CLINICAL TRIAL: NCT02663947
Title: Comparison of Optic Nerve Sheath Diameter Measured by Ultrasonography Before and After Ventriculoperitoneal Shunt Surgery in Adult Patients With Hydrocephalus
Status: Withdrawn | Type: Observational
Why Stopped: Because the investigator's workplace and department have been changed, this study cannot be carried out.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1091
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Hydrocephalus
Keywords: ventriculoperitoneal shunt; optic nerve sheath diameter; intracranial pressure
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasound group: ultrasonographic measure for optic nerve sheath diameter
  Interventions: Device: ultrasonographic measurement of optic nerve sheath diameter

INTERVENTIONS:
Device: ultrasonographic measurement of optic nerve sheath diameter — A thick layer of gel is applied on the upper closed eyelid. The linear 7.5-MHz ultrasound probe is then placed in the gel, without exerting pressure on the eye. Three measurements are taken for each optic nerve in the transverse plane, with the probe being horizontal. The final ONSD is the mean of these measurements.

SUMMARY:
Hydrocephalus is a disturbance of cerebrospinal fluid production, flow and absorption leading to intracranial hypertension. Assessment of the change in intracranial pressure after ventriculoperitoneal shunt surgery is important in guiding appropriate postoperative management. The optic nerve sheath diameter measured using ultrasonography has been verified as a non-invasive indicator of intracranial hypertension in various clinical studies. The investigators hypothesized that a change in optic nerve sheath diameter detected through ultrasonography could help ascertain a reduction in intracranial pressure following ventriculoperitoneal shunt surgery in adult patients without the risk of serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-90 years of age, ASA physical status 3 or less) who are scheduled for elective ventriculoperitoneal shunt surgery with non-communicating hydrocephalus and communicating hydrocephalus except for normal-pressure hydrocephalus
* Non-communicating hydrocephalus is defined as a pattern of ventricular system or at the level of the fourth ventricle's outlets by lesions including tumor, giant aneurysm, or aqueductal stenosis.
* Communicating hydrocephalus is defined as paraventricular enlargement resulting from postoperative complication after cranial surgery, meningitis, subarachnoid or intracerebral hemorrhage.

Exclusion Criteria:

* Patients with previous history of shunt operation, ocular disease and ocular surgery
* Patients with anatomical or functional abnormality of optic nerve
* emergency patient

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for elective ventriculoperitoneal shunt surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
ultrasonographic measurement of optic nerve sheath diameter | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Associate Professor Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019